CLINICAL TRIAL: NCT05981521
Title: Exploring the Association Between Paternal Age and Trisomy 21 Screening Results.
Brief Title: Paternal Age and Fetal Aneuploidy
Status: Completed | Type: Observational
Sponsor: Clinique Ovo (Industry)
Responsible Party: Sponsor
Other Study IDs: 3321
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Trisomy 21
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Optimo prenatal screening test — Prenatal screening test done between weeks 11 and 13 of pregnancy to detect conditions such as trisomy 13, 18 and 21

SUMMARY:
Trisomy 21, commonly known as down syndrome, is the most common chromosomal abnormality in humans. Advanced maternal age (AMA) is a well-recognized risk factor for trisomy 21, with the risk increasing significantly beyond the age of 35. Research on the effects of paternal age on the prenatal risk of trisomy 21 is lacking, with inconsistent findings in the literature.

The Harmony® prenatal test is an Non-Invasive Prenatal Testing (NIPT) that screens maternal blood for chromosomal abnormalities in the Cell-Free Fetal DNA (cfDNA). The harmony® prenatal test can detect conditions such as trisomy 13, 18, and 21, as well as sex chromosome abnormalities.

The Optimo test is a prenatal screening test that screens for trisomies 13, 18 and 21 in the developing fetus using extended biochemical screening in maternal. The Optimo test has shown high sensitivity and specificity in detecting trisomy 21.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18 years or older (at the time of trisomy 18 and 21 screening) and who were able to complete the questionnaire in either French or English
* Pregnant women who completed the entire trisomy 21 screening process at clinique ovo were included

Exclusion Criteria:

* Patients who did not indicate the male partner/donor's age were excluded
* Patients who did not complete or sign the clinical information form

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — We are evaluating genetic screening test on pregnant women.
Study Population: Pregnant women who underwent Optimo trisomy 21 screening at clinique ovo between January 2014 to June 2023
Sampling Method: Probability Sample
Enrollment: 7141 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Trisomy 21 screening results | 3 to 5 days
  On the day of the Optimo screening test, a questionnaire concerning clinical data (maternal and paternal age, ethnicity, weight, smoking status, pregnancy history) is completed. Blood test and nuchal transparency are done on that day. Results from serum analysis and nuchal transparency are combined to assess the risk of trisomy 21. Association between paternal age and trisomy 21 screening results will be assessed afterwards

CONTACTS AND LOCATIONS:
Overall Officials: Jacques I Kadoch, MD, Principal Investigator — clinique ovo R&D department
Locations (1):
- Clinique Ovo, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No